CLINICAL TRIAL: NCT06490835
Title: A Feasibility Study Protocol for Implementing Consultation-based Palliative Care Services to Provide High-quality Palliative Care to Families of Critically Ill Patients in Intensive Care Units: A Single-arm Pilot Study
Brief Title: Feasibility Study on Implementing Consultation-based High-quality Palliative Care Services in Intensive Care Units
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Shin Hye Yoo, Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2404-111-1532
Record Dates: First submitted 2024-06-24; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Critical Illness
Keywords: Intensive Care Units, Palliative Care, Decision Making
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Critically ill patients requiring ICU admission and their surrogates (Experimental): Participants receive high-quality palliative care through consultation-based palliative care services in addition to standard critical care.
  Interventions: Behavioral: High-quality palliative care through consultation-based palliative care services in the ICU

INTERVENTIONS:
Behavioral: High-quality palliative care through consultation-based palliative care services in the ICU — Family Counseling: Social workers implement a supportive process for families, assessing the individualized psychosocial and decisional support needs of patients and families to provide foundational data for palliative care consultations.
  Family Meeting Support: In cases of high medical complexity, uncertainty, value conflicts, or communication issues, the palliative care consultation team supports the facilitation of family meetings.
  Consultation: The palliative care team provides consultations to the attending physician based on the palliative care needs assessed during family counseling. Topics include symptom management, understanding treatment options, decisional conflict, emotional and practical support, goal of care setting, resources, and bereavement support.
  Palliative Care by attending Physician: The attending physician incorporates the consultations received from the palliative care consultation team to provide high-quality palliative care to patients and their families.

SUMMARY:
Critically ill patients in intensive care units (ICUs) receive life-sustaining treatments aimed at restoring or maintaining organ function. ICU admission often involves substantial physical and existential pressures that can burden patients, their families, and surrogates. Multidisciplinary palliative care support can help alleviate potential causes of suffering. Twenty patients admitted to the ICUs at Seoul National University Hospital, diagnosed with sudden and severe acute brain injury or progressive organ failure, along with their surrogates, will be enrolled in the study. This study aims to assess the feasibility of applying consultation-based palliative care services to provide higher quality palliative care for critically ill patients with acute illnesses and their families facing poor prognoses upon ICU admission. Additionally, the study seeks to determine whether providing such palliative care services can help better respect the patient's values and goals, reduce communication conflicts, alleviate family caregivers' anxiety and depression, and enhance satisfaction with critical care.

ELIGIBILITY:
Both patients and surrogates must meet the inclusion criteria and not fall under any exclusion criteria

[Inclusion Criteria]

Patients:

1. Diagnosis of sudden and severe acute brain injury due to at least one of the following etiologies: vascular, traumatic, metabolic, toxic, infectious, or anoxic AND
2. Glasgow Coma Scale score of 3-8 for at least 24 hours after the patient's admission AND
3. Unable to express themselves verbally or otherwise

OR

1. Diagnosis of advanced stage organ failure (any of the following)

   * Chronic lung disease requiring long-term oxygen therapy or mechanical ventilation
   * Decompensated liver cirrhosis
   * Chronic heart failure with NYHA class III or IV
   * Progressive neurological disease with a modified Rankin score of 3-5 (e.g., dementia, Parkinson's disease, and amyotrophic lateral sclerosis)
   * Three or more chronic comorbidities causing limitations in activities of daily living (ADL) AND
2. APACHE II score ≥ 14 at the time of screening AND
3. ICU stay of 7 days or more

Surrogates:

1. Family caregiver of a patient who meets the inclusion criteria (Family: defined as the patient's spouse, lineal ascendants and descendants within two degrees of kinship and their spouses, siblings and their spouses, and relatives within eight degrees of kinship and their spouses)
2. Aged 19 or older
3. Willing and able to provide consent for participation in the study

[Exclusion Criteria]

Patients:

1. Under 19 years of age
2. Unable to speak, understand, or read Korean
3. Refusal of palliative care consultation
4. Referred to palliative care prior to study enrollment
5. Within 48 hours of ICU admission
6. Presence of active cancer under treatment within 6 months prior to ICU admission
7. Care goals set to "comfort care" at the time of study enrollment
8. Death expected within 48 hours at the time of study enrollment
9. Lack of capacity to participate in the study without an appropriate surrogate

Surrogates:

1. Under 19 years of age
2. Unable to speak, understand, or read Korean
3. Determined by a physician to be in extremely poor health, making participation in the study infeasible
4. Refusal of palliative care consultation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Applying Consultation-Based High-Quality Palliative Care | 1 day (at discharge)
  Proportion of eligible contacts who consented and participated in the study, palliative care family counseling rate, and study completion rate.

SECONDARY OUTCOMES:
Change in Surrogates' Decisional Conflict before and after the Intervention | Pre-post comparison (baseline vs. within one week after consultation)
  The Decisional Conflict Scale (DCS) is a validated tool designed to evaluate personal uncertainty when making healthcare decisions, including modifiable factors that contribute to such uncertainty and the overall quality of the decision. It consists of 16 questions, each rated on a 5-point scale from "strongly agree" (1) to "strongly disagree" (5). Scores range from 16 to 80, with higher scores reflecting greater uncertainty and less favorable outcomes.
Change in Surrogates' Decisional Self-Efficacy before and after the Intervention | Pre-post comparison (baseline vs. within one week after consultation)
  The Decisional Self-Efficacy Scale (DSES) evaluates an individual's self-confidence or belief in their decision-making abilities, including the ability to participate in shared decision making. The scale consists of 11 items, each rated on a five-point Likert scale from "0" (no confidence) to "4" (very confident). To determine the total score, the sum of the item scores is divided by 11 and then multiplied by 25. Scores range between 0 and 100, with higher scores indicating higher levels of decision-making self-efficacy.
Change in Surrogates' Emotional State before and after the Intervention | Pre-post comparison (baseline vs. within one week after consultation)
  The Hospital Anxiety and Depression Scale (HADS) is a questionnaire consisting of fourteen items. Seven items focus on anxiety, while the other seven address depression. Scores for each subscale range from 0 to 21, with higher scores reflecting higher levels of anxiety or depression.
Surrogates' Decision Regret after the Intervention | Follow-up (within one week after consultation and one month after consultation; up to three months after the final consultation for deceased patients)
  The Decision Regret Scale (DRS) is a 5-item, 5-point Likert-type self-report measure used to assess distress or remorse following a healthcare decision. Items are rated from 1 ("strongly agree") to 5 ("strongly disagree"), with two items (2 and 4) phrased negatively. To calculate the total score, the negatively phrased items are first reversed, then the mean of all five items is computed. This mean is rescaled from 0 to 100 by subtracting 1 and multiplying by 25. A score of 0 represents no regret, while 100 indicates a high level of regret.
Level of Patient- and Family-Centered Care Experienced by Surrogates after the Intervention | Follow-up (within one week after consultation and one month after consultation; up to three months after the final consultation for deceased patients)
  The Modified Patient Perception of Patient-Centeredness (PPPC) scale, utilized by surrogates, consists of 12 items. The scores range from 0 to 100, with higher scores indicating a higher level of patient-centered care.
Surrogates' Satisfaction with the Intervention Services | Within one week after the final consultation
  Overall satisfaction with ICU palliative care, family counseling satisfaction, consultation satisfaction, and family meeting satisfaction, assessed on a 5-point scale (very dissatisfied, dissatisfied, neutral, satisfied, very satisfied)
Length of Hospital Stay | 1 day (at discharge)
  Length of ICU stay and overall hospital stay
Survival to Discharge Rate | 1 day (at discharge)
  Vital status at discharge
Days of Symptom Relief Treatments received in the ICU | 1 day (at discharge)
  Number of days receiving comfort-focused care (opioids and/or antipsychotics) during the ICU stay, based on a retrospective review of medical records
Proportion of Patients receiving Symptom Relief Treatments During the ICU stay | 1 day (at discharge)
  The percentage of the total study population who received comfort-focused care (opioids and/or antipsychotics) during the ICU stay, based on a retrospective review of medical records
Use of Life-Sustaining Procedures within 48 Hours before Death | 1 day (at discharge)
  We assessed the life-sustaining procedures administered during the end-of-life (EOL) stage using seven indicators: cardiopulmonary resuscitation (CPR), mechanical ventilation, continuous renal replacement therapy, surgery, vasopressors, extracorporeal membrane oxygenation (ECMO), and high-flow oxygen (HFO2). The percentage of the total study population that received each procedure within the last 48 hours of life was measured.
Use of Symptom Relief Treatments within 48 Hours before Death | 1 day (at discharge)
  Administration of opioid analgesics and/or antipsychotic medications within the final 48 hours of life was regarded as receiving end-of-life comfort care. We analyzed the percentage of the total study population that received opioid analgesics and/or antipsychotic medications during the last 48 hours of life.
Data Collection Completion Rate | Within three months after the final consultation
  Proportion of data collected at each time point exceeding 90%
Time Taken to Recruit Patients | Within the first year of study initiation
  Time interval between enrollment of the first and tenth patients

OTHER OUTCOMES:
Qualitative Evaluation of Intervention Feasibility and Satisfaction | Within three months after the final consultation
  Evaluation of feasibility and satisfaction through semi-structured, one-on-one interviews with surrogates
Additional Analysis of Surrogates' Emotional State Changes before and after the Intervention | One month after the final consultation (within three months for deceased patients)
  The Hospital Anxiety and Depression Scale (HADS) comprises fourteen questionnaire items, with seven dedicated to anxiety and the remaining seven to depression. Each subscale score ranges from 0 to 21, where higher scores indicate greater levels of anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Shin Hye Yoo, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, N/A (Not Applicable), South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeung YS, Kim Y, Kim S, Jung YS, Kim TJ, Yoo SH. Feasibility study protocol: implementing consultation-based high-quality palliative care services in intensive care units. BMJ Open. 2025 May 28;15(5):e093558. doi: 10.1136/bmjopen-2024-093558. PMID 40441768